CLINICAL TRIAL: NCT00003213
Title: A Randomized, Double-Blind Trial to Compare the Clinical Efficacy and Safety of Granisetron vs. Metoclopramide Combined to Dexamethasone in the Prophylaxis of Chemotherapy-Induced Delayed Emesis
Brief Title: Drugs to Reduce the Side Effects of Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SAKK 90/95; SWS-SAKK-90/95; EU-97035; CDR0000066073
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; nausea and vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Dexamethasone; dexamethasone acetate; Granisetron; Metoclopramide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Granisetron + Dexamethasone (Experimental): 1 mg Granisetron in the morning
  1 Metoclopramide placebo in the afternoon
  1 mg Granisetron in the evening 4 mg Dexamethasone in the morning
  Interventions: Drug: dexamethasone; Drug: granisetron hydrochloride
- Metoclopramide + Dexamethasone (Experimental): 20 mg Metoclopramide (1 x morning, 1 x afternoon, 1 x evening) 4 mg Dexamethasone in the morning
  Interventions: Drug: dexamethasone; Drug: metoclopramide hydrochloride

INTERVENTIONS:
Drug: dexamethasone — 4 mg Dexamethasone in the morning
  Other Names: dexamethasone acetate
Drug: granisetron hydrochloride — 1 mg Granisetron in the morning
  Other Names: Kytril®
  Arms: Oral Granisetron + Dexamethasone
Drug: metoclopramide hydrochloride — 20 mg Metoclopramide (1 x morning, 1 x afternoon, 1 x evening)
  Other Names: Metozolv®
  Arms: Metoclopramide + Dexamethasone

SUMMARY:
RATIONALE: Antiemetic drugs may help to reduce or prevent nausea and vomiting in patients treated with chemotherapy. It is not known whether receiving dexamethasone with granisetron is more effective than receiving dexamethasone with metoclopramide for reducing the side effects of chemotherapy.

PURPOSE: Randomized phase III trial to compare the effectiveness of dexamethasone with either granisetron or metoclopramide in patients treated with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the clinical efficacy and safety of Granisetron or Metoclopramide in combination with Dexamethasone in the prophylaxis of delayed nausea and vomiting induced by emetogenic cancer chemotherapy in patients with or without emesis in the acute phase.

OUTLINE: This is a randomized, double blind study. Patients are stratified by prior chemotherapy (yes vs no), regular alcohol consumption (yes vs no), and prior chemotherapy regimen (cisplatin/carboplatin vs others). Patients receive dexamethasone and granisetron by mouth bid on day 0. Patients are then randomized to receive either granisetron or metoclopramide with dexamethasone concurrently with chemotherapy. Arm I: Patients receive granisetron by mouth bid on days 1-5. Dexamethasone and a placebo are administered by mouth once daily on days 1-5. Arm II: Patients receive metoclopramide by mouth tid on days 1-5. Dexamethasone is administered by mouth once daily on days 1-5. Patients must complete a diary card daily for 6 days.

PROJECTED ACCRUAL: This study will accrue 360 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Scheduled to receive a first course of highly emetogenic single day cancer chemotherapy regimens including: Cisplatin at least 50 mg/m2 Carboplatin at least 300 mg/m2 Dacarbazine at least 500 mg/m2 Doxorubicin at least 40 mg/m2 Epirubicin at least 60 mg/m2 Ifosfamide at least 1200 mg/m2 Cyclophosphamide at least 600 mg/m2

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Must be able to complete diary card (fluent in German, French, or Italian) No severe concurrent illness No other etiologies that cause vomiting, including: Gastrointestinal obstruction Hypercalcemia CNS metastases No active peptic ulceration No prior gastrointestinal bleeding due to peptic ulcer No moderate to severe nausea or any vomiting in the 24 hours prior to chemotherapy Not pregnant or lactating

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 months since prior chemotherapy Concurrent etoposide and fluorouracil allowed (days 1-5) No chemotherapy before day 0 of study Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No other concurrent antiemetics No concurrent high dose benzodiazepines No concurrent psychotropic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 1996-05; Primary Completion 1999-04 (Actual); Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Complete and partial control of emesis | Total control of emesis on every one of the 5 days following the acute phase

CONTACTS AND LOCATIONS:
Overall Officials: Matti S. Aapro, MD, Study Chair — European Institute of Oncology
Locations (10):
- Istituto Europeo Di Oncologia, Milan, Italy
- Switzerland (9):
  - Kantonspital Aarau, Aarau
  - Office of Walter Weber-Stadelman, Basel
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Hopital Cantonal Universitaire de Geneva, Geneva
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Burgerspital, Solothurn, Solothurn
  - City Hospital Triemli, Zurich
  - Klinik Hirslanden, Zurich

REFERENCES:
- [Result] Aapro MS, Thuerlimann B, Sessa C, De Pree C, Bernhard J, Maibach R; Swiss Group for Clinical Cancer Research. A randomized double-blind trial to compare the clinical efficacy of granisetron with metoclopramide, both combined with dexamethasone in the prophylaxis of chemotherapy-induced delayed emesis. Ann Oncol. 2003 Feb;14(2):291-7. doi: 10.1093/annonc/mdg075. PMID 12562658
- [Result] Bernhard J, Maibach R, Thurlimann B, Sessa C, Aapro MS; Swiss Group for Clinical Cancer Research. Patients' estimation of overall treatment burden: why not ask the obvious? J Clin Oncol. 2002 Jan 1;20(1):65-72. doi: 10.1200/JCO.2002.20.1.65. PMID 11773155